CLINICAL TRIAL: NCT05005156
Title: A Phase IIb Clinical Trial to Evaluate the Efficacy, Safety and Immunogenicity of Two Doses of Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) in Adults 18 Years of Age and Older, Living With HIV.
Brief Title: Phase IIb Trial of Recombinant Novel Coronavirus Vaccine (Ad5-nCoV) in Adults 18 Years of Age and Older, Living With HIV
Acronym: COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Huésped (Other)
Collaborators: Canadian Center for Vaccinology (Other); CanSino Biologics Inc. (Industry); Hospital Fernandez (Other)
Responsible Party: Principal Investigator, Pedro Cahn, Scientific Director, MD; PhD, Fundación Huésped
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FH-58
Record Dates: First submitted 2021-06-07; First posted 2021-08-13 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Covid19
Keywords: Adenovirus 5, HIV, COVID19, vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This Phase IIb study is a clinical trial for 500 participants 18 years of age or older living with HIV. All participants will receive two doses of the study vaccine and will be followed to monitor vaccine candidate safety, immunogenicity, and efficacy during 52 weeks. Fifty five days after the first vaccination, all participants will receive a second injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active vaccine Ad5-nCoV (Experimental): Active vaccine Ad5-nCoV, 0.5 mL/vial
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) (Ad5-nCoV)
- Placebo for Ad5-nCoV (Placebo Comparator): Placebo for Ad5-nCoV, 0.5 mL/vial
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) (Ad5-nCoV)

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) (Ad5-nCoV) — All participants will receive two doses vaccine and will be followed to monitor vaccine candidate safety, immunogenicity, and efficacy for a duration of 52 weeks. Fifty four days after the first vaccination, all participants will receive a second injection.

SUMMARY:
A randomized, double-blind, placebo -controlled, phase IIb clinical trial to evaluate the efficacy, safety and immunogenicity of one or two doses of Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) in adults 18 years of age and older, living with HIV, on stable treatment, and virologically suppressed for at least 6 months

Protocol number: FH-58

DETAILED DESCRIPTION:
Primary Safety Objectives:

* Evaluate the incidence of solicited adverse reactions within 7 days after vaccination.
* Evaluate the incidence of unsolicited adverse events within 28 days after vaccination.
* Evaluate the HIV viral load 24 and 52 weeks after vaccination
* Evaluate the incidence of serious adverse events (SAE) and medically attended adverse events (MAE) within 52 weeks after vaccination in all participants.

Primary Immunogenicity Objectives:

* Evaluate the seroconversion rate of S-RBD IgG antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination, measured by ELISA.
* Evaluate the immunogenicity of two doses of the vaccine.

Secondary Safety Objectives:

* Evaluate the incidence of a decrease in CD4+ cell count by ≥20% at 24 and 52 weeks after vaccination.
* Evaluate changes in the CD4/CD8 ratio at 24 and 52 weeks compared to the basal value.
* To evaluate the efficacy of two doses of Ad5-nCoV in different age groups from 14 and 28 days to 24 and 52 weeks after vaccination. This will be evaluated by weekly participant contact to assess for any signs or symptoms of COVID 19.

Secondary Immunogenicity Objectives:

* Evaluate the GMT of S-RBD IgG antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination, measured by ELISA.
* Evaluate the GMI of S-RBD IgG antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination, measured by ELISA.
* Evaluate the seroconversion rate of pseudo-virus neutralizing antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination.
* Evaluate the GMT of pseudo-virus neutralizing antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination.
* Evaluate the GMI of pseudo-virus neutralizing antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination.
* Evaluate the positive rate and level of IFN-γ, TNF, IL-4, IL-5, IL-13 stimulated by peptide pool of S protein on Day 28, Day 84 and Weeks 24 and Week 52 after vaccination, measured by intracellular cytokine staining (ICS) (in a subset of approximately 50 participants).

Exploratory Objectives

* To evaluate the efficacy of two doses of Ad5-nCoV in preventing virologically confirmed (PCR positive) COVID-19 disease occurring 14 days and 28 days to 52 weeks after vaccination, regardless of severity.
* To evaluate the efficacy of two doses of Ad5-nCoV in preventing virologically (PCR) or serologically (four-fold increase in SARS-CoV-2 anti-N IgG from pre-immunization to post symptom, defined as Day 21-28 post illness blood test, or pre-symptom to post-symptom blood test) confirmed COVID-19 disease occurring 14 and 28 days to 52 weeks after vaccination, regardless of severity.
* To evaluate the efficacy of two doses of Ad5-nCoV in preventing severe COVID-19 disease caused by SARS-CoV-2 infection from 14 and 28 days to 24 and 52 weeks after vaccination.

Severe disease is defined as: 1) Clinical signs at rest indicative of severe systemic illness (respiratory rate ≥ 30 per minute, heart rate ≥ 125 per minute, SpO2 ≤ 93% on room air at sea level or PaO2/FiO2 < 300 mm Hg), 2) Respiratory failure (defined as needing high-flow oxygen, non-invasive ventilation, mechanical ventilation or ECMO), 3) Evidence of shock (SBP < 90 mm Hg, DBP < 60 mm Hg, or requiring vasopressors), 4) Significant acute renal, hepatic, or neurologic dysfunction, 5) Admission to an ICU

* Evaluate the efficacy of Ad5-nCoV in preventing asymptomatic disease of COVID-19 (confirmed by N IgG antibody on week 52 after vaccination).
* Evaluate the severity of COVID-19 cases among vaccine recipients (based on WHO or FDA criteria) as compared to the control group, to measure antibody-mediated disease enhancement (ADE).
* Evaluate for any evidence of SARS-CoV-2 virus shedding in COVID-19 cases that occurred 28 days to 52 weeks after vaccination (detection of viral nucleic acid every 2 days after being confirmed).
* Perform genotyping of SARS-CoV-2 virus isolates of COVID-19 cases that occurred 28 days to 52 weeks after vaccination.
* Evaluate incidence of suspected but unconfirmed cases of COVID-19 (either because of negative or no tests).

ELIGIBILITY:
Inclusion Criteria:

1. Adults of 18 years of age, and older.
2. Confirmed HIV infection

   * At least two HIV plasma viral load (pVL) below 40 copies in the last 12 months, one within the last 60 days (value obtained at Screening visit can be used for the value within the last 60 days)
   * A CD4 count at screening equal or above 300 cells/mL and a CD4 percentage equal or above 15 % within the previous 60 days (value obtained at Screening visit can be used for the value within the last 60 days)
   * Participant must be on a stable highly active anti-retroviral treatment (HAART) for 6 months (unless the change is due to tolerability, in which case the regimen can be for only the previous 3 months) and with an estimated adherence of ≥80% within the last 60 days. - A HAART regimen (as defined by the Argentinean ART guidelines), means a combination of 2 NRTIs plus one INSTI or a NNRTI or a boosted PI or a dual combination of dolutegravir and 3TC.
3. Able and willing (in the Investigator's opinion) to comply with all study requirements.
4. Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner/personal doctor and access all medical records when relevant to study procedures.
5. Healthy adults, or stable-healthy adults who may have a pre-existing medical condition that does not meet any exclusion criteria. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
6. For females of childbearing potential only, willingness to practice continuous effective contraception (see glossary) for 30 days prior to enrollment in the study, for 90 days after receiving vaccination during the study, and have a negative pregnancy test on the day(s) of screening/ vaccination (First Injection Visit and Second Injection Visit).
7. Males participating in this study who are involved in heterosexual sexual activity must agree to practice adequate contraception (see glossary) and refrain from donating sperm for 90 days after receiving the study vaccination.
8. Agreement to refrain from blood donation during the study.
9. Provide written informed consent.

Exclusion Criteria:

* 1. Participation in any other COVID-19 prophylactic drug trials for the duration of the study.

Note: Participation in COVID-19 treatment trials is allowed in the event of hospitalization due to COVID-19. The study team should be informed as soon as possible. 2. Participation in SARS-CoV-2 serological surveys where participants are informed of their serostatus for the duration of the study.

Note: Disclosure of serostatus post enrolment may accidentally unblind participants to group allocation. Participation in this trial can only be allowed if volunteers are kept blinded to their serology results from local/national serological surveys 3. Planned receipt of any vaccine (licensed or investigational), other than the study intervention, within 14 days before and after study vaccination 4. Prior receipt of an investigational or licensed vaccine likely to impact on the interpretation of the trial data (e.g. Adenovirus vectored vaccines, any coronavirus or SARS vaccines) 5. Administration of immunoglobulins and/or any blood products within the three months prior to the planned administration of the vaccine candidate 6. Any confirmed or suspected immunosuppressive or immunodeficient state (other than living with HIV, on stable treatment, and virologically suppressed for at least 6 months); asplenia; recurrent severe infections and chronic use (more than 14 days) of immunosuppressant medication within the past 6 months. Topical steroids or short-term (course lasting ≤14 days) oral steroids are not an exclusion 7. Active opportunistic infections or other AIDS-defining illness in the last six months.

8. History of allergic disease or reactions likely to be exacerbated by any component of Ad5-nCoV 9. Any history of angioedema 10. Any history of anaphylaxis to any vaccine component 11. Pregnancy, lactation or willingness/intention to become pregnant within 90 days after receiving study vaccine 12. Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ) 13. History of serious psychiatric condition likely to affect participation in the study 14. Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture 15. Suspected or known current alcohol or drug dependency 16. Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness (mild/moderate well-controlled comorbidities are allowed) 17. History of laboratory-confirmed COVID-19 18. Continuous use of anticoagulants, such as coumarins and related anticoagulants (i.e. warfarin) or novel oral anticoagulants (i.e. apixaban, rivaroxaban, dabigatran and edoxaban) 19. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Evaluate the incidence of solicited adverse reactions at 7 days after vaccination | 7 days after vaccine
  Evaluate the incidence of solicited adverse reactions at 7 days after vaccination
Evaluate the incidence of unsolicited adverse events at 28 days after vaccination | 28 days after vaccine
  Evaluate the incidence of unsolicited adverse events at 28 days after vaccination
Suppression of HIV viral load at 24 and 52 weeks | 52 weeks after vaccination
  Percentage of suppressed HIV viral load
Evaluate the incidence of serious adverse events (SAE) and medically attended adverse events | 52 weeks after vaccination in all participants.
  Evaluate the incidence of serious adverse events (SAE) and medically attended adverse events events (MAE)
Evaluate the antibody response attended adverse | during 52 weeks after vaccination
  ● Evaluate the seroconversion rate of S-RBD IgG antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination, measured by ELISA.
Compare antibody response in both group | during 52 weeks after vaccination
  compare the seroconversion rate of S-RBD IgG antibody of one dose versus two doses of the vacccine

SECONDARY OUTCOMES:
Evaluate impact in CD4* cell | during 52 weeks after vaccination
  Evaluate the incidence of a decrease in CD4+ cell count by ≥20%
Evaluate impact in ratio CD4/CD8 | during 52 weeks after vaccination
  Evaluate changes in the CD4/CD8 ratio at 24 and 52 weeks compared to the basal value.
Geometric mean antibody titers | during 52 weeks after vaccination
  ● Evaluate the GMT of S-RBD IgG antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination, measured by ELISA
Geometric Mean Increase | during 52 weeks after vaccination
  Evaluate the GMI of S-RBD IgG antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination, measured by ELISA.
Evaluate the seroconversion rate of pseudo-virus neutralizing antibody | during 52 weeks after vaccination
  Evaluate the GMT and GMI of pseudo-virus neutralizing antibody on Day 28, Day 84 and Week 24 and Week 52 after vaccination.
Evaluate impact in chemokines | during 52 weeks after vaccination
  Evaluate the positive rate and level of IFN-γ, TNF, IL-4, IL-5, IL-13 stimulated by peptide pool of S protein measured by intracellular cytokine staining (ICS) (in a subset of approximately 60 participants).

OTHER OUTCOMES:
Evaluate impact in preventing CoVID-19 confirmed cases | from 14 days after vaccination
  o evaluate the efficacy of one or two doses of Ad5-nCoV in preventing virologically (PCR) or serologically (four-fold increase in SARS-CoV-2 anti-N IgG from preimmunization to post symptom, defined as Day 21-28 post illness blood test, or presymptom to post-symptom blood test) confirmed COVID-19 disease, regardless of severity confirmed (PCR positive) COVID-19 disease, regardless of severity
Identify variants of interest and concern | during 52 weeks after vaccination
  Perform genotyping of SARS-CoV-2 virus isolates of COVID-19 cases
Evaluate the incidence of CoVID19 confirmed by IgG antibody disease of COVID-19 confirmed by N IgG antibody | week 52 after vaccination
  Evaluate the efficacy of one or two doses of Ad5-nCoV in asymptomatic disease of COVID-19 confirmed by N IgG antibody
Evaluate the severity of COVID-19 cases | week 52 after vaccination
  Evaluate the severity of COVID-19 cases among vaccine recipients (based on WHO or FDA criteria) as compared to the control group, to measure antibody-mediated disease enhancement
Evaluate incidence of suspected but unconfirmed cases of COVID-19 (either because of negative or no tests). | week 52 after vaccination
  Evaluate incidence of suspected but unconfirmed cases of COVID-19 (either because of negative or no tests).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Cahn, MD:PhD, Principal Investigator — fundacion huesped
Locations (4):
- Argentina (4):
  - Fundacion Huesped, CABA, Buenos Aires
  - Centro de Estudio Infectologicos (CEI), Capital Federal, Buenos Aires
  - Helios Salud, Capital Federal, Buenos Aires
  - Hospital Fernandez, Capital Federal, Buenos Aires

REFERENCES:
- [Derived] Cahn P, Barreto L, Figueroa MI, Fink V, Rolon MJ, Lopardo G, Cassetti I, Ceschel M, Patterson P, Gambardella L, Mernies G, Nava A, Gou J, Wang R, Zhu T, Halperin SA. Immune response induced by the recombinant novel coronavirus vaccine (Adenovirus type 5 vector) (Ad5-nCoV) in persons living with HIV (PLWH). PLoS One. 2025 Jun 11;20(6):e0312893. doi: 10.1371/journal.pone.0312893. eCollection 2025. PMID 40498774

DOCUMENTS (1):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT05005156/Prot_000.pdf